CLINICAL TRIAL: NCT02917564
Title: Subtenons Triamcinolone Acetonide Injections for Treatment of Persistent Choroidal Effusions Post Glaucoma Surgery
Brief Title: Triamcinolone Injections for Persistent Choroidal Effusions Post Glaucoma Surgery
Acronym: TRICEPS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Catherine Birt, Ophthalmologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 474-2015
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Glaucoma; Choroidal Effusions
Keywords: Choroidal effusions; Trabeculectomy
MeSH Terms: conditions — Glaucoma; Choroidal Effusions | interventions — Triamcinolone Acetonide; Suspensions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Patients placed in a semi supine position. A cotton-tipped applicator saturated with proparacaine 0.5% (Alcaine, Alcon Labs) is placed into the conjunctival fornix of the supero-temporal quadrant for 5 minutes following initial proparacaine drops.
  After anaesthetic medication is placed, a 3 ml syringe will be placed into the superotemporal conjunctival fornix but no needle is present and no drug injected.
  Interventions: Other: Sham - Participants will not recieve the Triamcinolone Acetonide
- Injection (Active Comparator): Patients placed in a semi supine position. A cotton-tipped applicator saturated with proparacaine 0.5% (Alcaine, Alcon Labs) is placed into the conjunctival fornix of the supero-temporal quadrant for 5 minutes following initial proparacaine drops.
  After anaesthetic medication is placed, 1mL of a 40 mg/ml suspension of triamcinolone acetonide is injected through the superotemporal conjunctival fornix using a 25 Gauge needle, 5/8 inch length on a 3 ml syringe, following the contour of the globe with the needle, external to sclera for the full length of the needle such that the needle tip is ultimately positioned immediately posterior to the macula with the bevel down.
  Interventions: Drug: Triamcinolone Acetonide 1 ml of 40 mg/mL suspension

INTERVENTIONS:
Drug: Triamcinolone Acetonide 1 ml of 40 mg/mL suspension — After preparation, Triamcinolone Acetonide 1 ml of 40 mg/mL suspension is injected through the superotemporal conjunctival fornix using a 25 Gauge needle, 5/8 inch length on a 3 ml syringe, following the contour of the globe with the needle, external to sclera for the full length of the needle such that the needle tip is ultimately positioned immediately posterior to the macula with the bevel down.
  Other Names: Kenalog
  Arms: Injection
Other: Sham - Participants will not recieve the Triamcinolone Acetonide — Patients will be given a sham.
  Arms: Control

SUMMARY:
During glaucoma surgery, a new opening is created that allows fluid to drain out of the eye, bypassing the clogged drainage channels that are malfunctioning in patients with glaucoma. In some patients who have had glaucoma surgery too much fluid flows out and this results in a pressure that is too low. This may cause swelling of one layer at the back of the eye called the choroid. The formation of this swelling, called a choroidal effusion or "choroidal", often makes the eye pressure stay too low, and one of the results is a decrease in vision. The treatment for a choroidal effusion is to try to raise the eye pressure somewhat to allow the swelling to subside. In our clinical work, we have found that an injection with an anti-inflammatory drug called triamcinolone appears to be helpful in speeding up healing. We plan to compare two groups of patients with choroidal effusions, one group that gets an injection of triamcinolone and one that gets a "sham" treatment with nothing injected and compare the length of time it takes the choroidal effusions to disappear. Both groups receive the standard treatment with eye drops. We will also assess the outcome of the glaucoma surgery and any other complications that may occur. This research is aimed at studying a new method of improving the outcomes of surgery for glaucoma patients, and further the treatment of glaucoma.

DETAILED DESCRIPTION:
Glaucoma is the second commonest cause of blindness in our society. The only effective treatment currently involves lowering the intraocular pressure (IOP) by medical, laser, or surgical techniques. Glaucoma surgery is indicated when further IOP lowering is needed despite maximal medical therapy and appropriate laser treatment.

The choroid is a pigmented and vascular structure located between the sclera and retinal pigmented epithelium.

Choroidal effusions are aberrant collections of fluid within the suprachoroidal potential space. There are two types of choroidal effusion, serous and hemorrhagic, depending on the type of fluid that accumulates in the suprachoroidal space. A serous choroidal effusion is composed of a transudate fluid from increased transmural pressure across the capillaries. Their development is usually relatively painless. Hemorrhagic choroidal effusion or suprachoroidal haemorrhage is a sudden and usually very painful accumulation of blood in the suprachoroidal space. 4 Choroidal effusions can be caused by both low IOP and pro-inflammatory conditions. Causes of concomitant low IOP and inflammation include trauma and eye surgery, especially glaucoma surgery. Inflammatory causes include scleritis.

Modern glaucoma surgery has minimized the incidence of postoperative hypotony and resultant choroidal effusion but it is still prevalent. 1 The prevalence of choroidal effusions after glaucoma surgery varies between 10 and 15%, with average of 13% after trabeculectomy (the standard technique of glaucoma surgery). 5 A complication of low-IOP-induced choroidal effusion is hypotony maculopathy, which can cause permanent decline in vision, especially if not resolved in a timely manner. 5 Treatment can be either medical or surgical. Medical treatment includes cessation of any systemic and topical IOP lowering agents and adding cycloplegic agents, topical steroids and eventually systemic steroids. If treatments do not increase the IOP and reduce the choroidal effusion, then surgical management should be considered.

Depending on the particular clinical circumstances of each patient, different surgical approaches can be used, including revision of the trabeculectomy flap, anterior chamber reformation, and surgical drainage of the effusion.

As an alternative to systemic steroids, steroids as triamcinolone acetonide (Kenalog™) can be injected in the subtenons space. This treatment allows for a high local dose of steroids, without exposing the patient to systemic treatment. Not every patient requires steroid injection, and this treatment will be reserved for patients who do not respond to medical management after a few days.

Following the sham or Kenalog injection participants will receive topical prednisolone acetate 1% qid for 4 weeks or PRN Topical atropine 1% qid for one week or PRN.

There are several studies in the literature showing the benefit of a triamcinolone injection for different inflammatory conditions, such uveitis and for the treatment of diabetic maculopaty and cystoid macular edema. 6-9 Recently Shen et al. published the benefit of subtenons triamcinolone acetonide in the management of a combination of retinal detachment and choroidal effusion. 2 However we did not find any studies that assessed the benefit on triamcinolone subtenons injection for choroidal effusion after glaucoma surgery. In a recent retrospective study we performed a chart review of the effect of subtenons triamcinolone injection in patients with choroidal effusions after glaucoma surgery compared to a group of patients who did not receive the injection as part of their management. We found that recovery time in the injection group was significantly shorter than in patients with no injection, 10.6 days versus 27.44 days. (p=0.02). The study showed no difference in final intraocular pressure (IOP), number of medications and visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Patients who have had glaucoma surgery at Sunnybrook Health Sciences Centre and / or Kensington Eye Institute and developed choroidal effusions that do not improve after one week of standard medical treatment. (Trabeculectomy, Combined Phaco-trabeculectomy, Glaucoma tube Shunts, postoperative 5-FU needling, and laser suture lysis are all considered as eligible Glaucoma surgeries/Procedures)
* Decision makers fluent in English.
* Decision makers able to understand and read consent form.

Exclusion Criteria:

* Patients with choroidal effusions with improvement after one week of medical treatment.
* Patients with choroidal hemorrhage, demonstrated clinically and or with B Scan.
* Patients with aqueous misdirection and IOP > 10 mmHg.
* Patients that refuse subtenons injection.
* Patients with signs of infection.
* Patients with choroidal effusions who did not have glaucoma surgery.
* Patients unable to follow up within study schedule.
* Female patients of childbearing potential who are pregnant of do not agree to use adequate methods of contraception from time of enrollment until 40 days after the last day of Triamcinolone administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to resolution | One week to three months
  The time to clinical resolution of the choroidal effusions will be determined

SECONDARY OUTCOMES:
IOP | 3 month visit
  Intraocular pressure at the final study visit
Vision | 3 month visit
  Visual acuity at the final study visit
Medications | 3 month visit
  Number of glaucoma medications required at the final study visit
Complications | All study visits
  Any intra-operative or post-procedural side effects or complications, including further surgery, will be recorded and compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Birt, MD FRCSC, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Summary data will be reported, individual participant data will not